CLINICAL TRIAL: NCT01061255
Title: Physiological and Psychological Responses to Stress in Year 6 Medical Students Faced to Ambulatory Symptomatic Patients
Brief Title: Stress and Clinical Reasoning in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BRD/09/08-M
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Stress
Keywords: Stress; Cortisol; Clinical reasoning; Ambulatory setting; Medical students; Year 6 medical students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluation of the stress — Medical Students having to solve a medical problem in ambulatory setting (studied group) vs. in hospitalisation setting (control group).
  Measures: The French version of the Anxiety Spielberger test is administered just before and after each problem solving session.
  Cortisol salivary samples are taken before and after each problem solving session. Salivary cortisol levels have been shown to be correlated to stressful situations and some personality traits but with some difference according to gender.

SUMMARY:
Solving a problem in ambulatory setting may contain peripheral stress due to socio-evaluative stressors (patient's expectations about explanations) and task contingent stress due to time pressure, the necessity to take into account patient's mood, to deal with uncertainty of their own data collection and with complex clinical situations. In France, excepted for family medicine, undergraduate medical students and residents are currently not trained to perform consultations and are never exposed to ambulatory patients during training. The investigators postulate that this lack of practice may generate a significant state of stress during the first consultations and consequently modify or even impair clinical reasoning.

The primary objective of this study is to compare subjective and physiological levels of acute stress in ambulatory versus hospitalization setting in medical students confronted to a real patient with a diagnostic problem.

Measures: The French version of the Anxiety Spielberger test is administered just before and after each problem solving session.

Cortisol salivary samples are taken before and after each problem solving session. Salivary cortisol levels have been shown to be correlated to stressful situations and some personality traits but with some difference according to gender.

Cognitive appraisal (threat/challenge) is assessed before and after the tasks by the ratio of primary appraisal to secondary appraisal according to Tomaka et al.

DETAILED DESCRIPTION:
Participants and Method:

Year 6 medical students who attend a one-month full-time course in an Internal Medicine Department are eligible.

Since no consultations in the ambulatory setting are currently structured for medical students, the following adjustments have been done within the internal medicine consultation department, with the approval of the department director:

* the consultation duration has been increased (1 hour instead of 30 minutes)
* during the first 30 minutes, consultation is performed by the participant
* during the following 30 minutes, the patient is examined by his/her own physician.
* The consent of the patient has been obtained by phone (prior to the consultation).

ELIGIBILITY:
Inclusion Criteria:

* Year 6 medical students who attend a one-month full-time course in an Internal Medicine Department

Exclusion Criteria:

* Student who repeats his year 6 of medicine
* Student treated with corticoids

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2010-04-12 (Actual); Study Completion 2010-04-12 (Actual)

PRIMARY OUTCOMES:
Increase in salivary cortisol and in Spielberger score | one hour

SECONDARY OUTCOMES:
Difference in the cognitive appraisal (challenge or threat) | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Pierre POTTIER, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France